CLINICAL TRIAL: NCT02372279
Title: Prospective Randomized Study to Evaluate the Effect of Embryonic Observation on the Live Birth Rate (LBR)
Brief Title: Prospective Randomized Study to Evaluate the Effect of Embryonic Observation on the Gestation (PROdE)
Acronym: PROdE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The forecast regarding the number of patients that could enter the study were not met in the designated period
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Jorge Ten Morro, Ph.D. Embryologist, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: InstitutoBernabeu
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Placenta; Implantation
Keywords: Embryo development; Implantation; In vitro fertilization

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No embryo observation (NEO) (No Intervention): Study group. No embryonic observation from day one to day five of embryo development.
- Embryo observation (EO) (Experimental): Control group. Conventional embryonic observations performed in day two, three and five of embryo development.
  Interventions: Other: Embryo observation

INTERVENTIONS:
Other: Embryo observation — In EO group, conventional observations will be made.
  Arms: Embryo observation (EO)

SUMMARY:
In a conventional in vitro fertilization (IVF) cycle, daily microscopic observation of embryos outside the incubator to assess their morphology and establish a selection process is performed. In this way it is possible to know which embryo or embryos have greater implantantion capacity and will be transferred to the uterus to obtain a viable pregnancy. However, these observations can produce deleterious effects on embryo development due to changes in temperature, pH and osmolarity of the culture media, as well as a negative effect of direct light microscope for observation. This project aims to test the hypothesis that non-embryonic observation produces a beneficial effect on embryo quality until day 5 of development (blastocyst stage) and, therefore, on rates of implantation and ongoing gestation, compared with the conventional protocol of observations under the inverted microscope on days two, three and five of development.

DETAILED DESCRIPTION:
The present study is a prospective double-blind randomised controlled trial (RCT) approved by a local Ethics Committe. Summarily, in the control group we did three embryo observations outside the incubator as we usually do in our conventional protocol: day 2, day 3 and day 5, just before ET; in the study group we performed a unique embryo observation on day 5 before ET. All the subjects that participated in the study were informed and gave us their consent to take part on it.

The inclusion criteria of the study were: first cycle of ART treatment with conventional IVF or ICSI with donated eggs, normal uterine cavity and a single or double embryo transfer, always performed on day 5 at blastocyst stage.

The exclusion criteria were the following: patients above 50 years old, patients that were diagnosed with recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL) or uterine pathologies, body mass index >30 kg/m2, the use of seminal samples coming from donors or testicular origin and cycles that included preimplantational genetic testing (PGT).

LBR was the main outcome of our study, defined as the number of deliveries that resulted in a live born neonate, expressed per 100 embryo transfers (Zegers- Hochschild et al., 2009). Secondary efficacy endpoints were positive hCG rate (>5 mUI/mL, assessed in serum 14 days after oocyte retrieval), implantation rate (number of gestational sacs observed divided by the number of embryos transferred, expressed as a percentage, %), ongoing pregnancy rate, defined as a pregnancy with a detectable heart rate at 12 weeks of gestation or beyond and miscarriage (loss of a pregnancy after 12 weeks of gestation).

In addition, we assessed the next IVF laboratory parameters: fertilization rate, blastocyst formation rate on day 5, blastocyst quality, number of transferred embryos and number of usable blastocysts (number of blastocysts transferred and frozen).

The sample size calculation was based on the primary outcome. We assumed a live birth rate of 40% in the control group, compared to 50% in the non-observational group deduced from previous studies. By applicating the sample size calculation program, 776 patients (388 per group) were required in order to detect a risk difference (RD) of 10% between the two groups in the final analysis, with a power of 80% at a two-sided, adjusted alpha-level of 0.05. A follow-up loss rate of 10% was estimated.

ELIGIBILITY:
Inclusion Criteria:

* First cycle of ART treatment with conventional IVF or ICSI with donated eggs.
* Normal uterine cavity and a single or double embryo transfer, always performed on day 5 at blastocyst stage.

Exclusion Criteria:

* Patients above 50 years old, patients that were diagnosed with recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL) or uterine pathologies,
* Body mass index >30 kg/m2.
* The use of seminal samples coming from donors or testicular origin.
* Cycles that included preimplantational genetic testing (PGT).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate | Nine months after treatment.
  The number of deliveries that resulted in a live born neonate, expressed per 100 embryos

SECONDARY OUTCOMES:
Positive hCG rate | 14 days after oocyte retrieval.
  Number of treatments with a level of BhCG >5 mUI/mL, assessed in serum.
Implantation rate | 6-7 weeks after oocyte retrieval.
  Number of gestational sacs observed divided by the number of embryos transferred. expressed as a percentage, %.
Ongoing pregnancy rate | 12 weeks after B-hCG positive test
  Defined as a pregnancy with a detectable heart rate at 12 weeks of gestation or beyond.
Miscarriage rate | From 12 weeks after gestation to delivery
  Loss of a pregnancy after 12 weeks of gestation.
Fertilization rate | 16-18 hours after microinjection or insemination
  Number of fertilized oocytes out of the total microinjected or inseminated.
Blastocyst formation rate on day 5 | 5 days after microinjection or insemination.
  Number of embryos that reach the blastocyst stage at day 5
Blastocyst quality | 5 days after microinjection or insemination.
  The assessment of blastocyst morphology in several grades
Number of usable blastocysts | 5 days after microinjection or insemination.
  Number of blastocysts transferred and frozen.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ten Morro, Ph.D., Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain

REFERENCES:
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182
- [Background] Fujiwara M, Takahashi K, Izuno M, Duan YR, Kazono M, Kimura F, Noda Y. Effect of micro-environment maintenance on embryo culture after in-vitro fertilization: comparison of top-load mini incubator and conventional front-load incubator. J Assist Reprod Genet. 2007 Jan;24(1):5-9. doi: 10.1007/s10815-006-9088-3. Epub 2006 Dec 13. PMID 17160731
- [Background] Gardner DK, Lane M, Stevens J, Schlenker T, Schoolcraft WB. Blastocyst score affects implantation and pregnancy outcome: towards a single blastocyst transfer. Fertil Steril. 2000 Jun;73(6):1155-8. doi: 10.1016/s0015-0282(00)00518-5. PMID 10856474
- [Background] Bernabeu R, Roca M, Torres A, Ten J. Indomethacin effect on implantation rates in oocyte recipients. Hum Reprod. 2006 Feb;21(2):364-9. doi: 10.1093/humrep/dei343. Epub 2005 Nov 10. PMID 16284067
- [Background] Herrero J, Tejera A, Albert C, Vidal C, de los Santos MJ, Meseguer M. A time to look back: analysis of morphokinetic characteristics of human embryo development. Fertil Steril. 2013 Dec;100(6):1602-9.e1-4. doi: 10.1016/j.fertnstert.2013.08.033. Epub 2013 Sep 29. PMID 24083877
- [Background] Zhang JQ, Li XL, Peng Y, Guo X, Heng BC, Tong GQ. Reduction in exposure of human embryos outside the incubator enhances embryo quality and blastulation rate. Reprod Biomed Online. 2010 Apr;20(4):510-5. doi: 10.1016/j.rbmo.2009.12.027. Epub 2009 Dec 28. PMID 20129824
- [Background] Kirkegaard K, Kesmodel US, Hindkjaer JJ, Ingerslev HJ. Time-lapse parameters as predictors of blastocyst development and pregnancy outcome in embryos from good prognosis patients: a prospective cohort study. Hum Reprod. 2013 Oct;28(10):2643-51. doi: 10.1093/humrep/det300. Epub 2013 Jul 30. PMID 23900207
- [Background] Steptoe PC, Edwards RG. Birth after the reimplantation of a human embryo. Lancet. 1978 Aug 12;2(8085):366. doi: 10.1016/s0140-6736(78)92957-4. No abstract available. PMID 79723
- [Background] Bognar Z, Csabai TJ, Pallinger E, Balassa T, Farkas N, Schmidt J, Gorgey E, Berta G, Szekeres-Bartho J, Bodis J. The effect of light exposure on the cleavage rate and implantation capacity of preimplantation murine embryos. J Reprod Immunol. 2019 Apr;132:21-28. doi: 10.1016/j.jri.2019.02.003. Epub 2019 Mar 4. PMID 30852462
- [Background] Barberet J, Chammas J, Bruno C, Valot E, Vuillemin C, Jonval L, Choux C, Sagot P, Soudry A, Fauque P. Randomized controlled trial comparing embryo culture in two incubator systems: G185 K-System versus EmbryoScope. Fertil Steril. 2018 Feb;109(2):302-309.e1. doi: 10.1016/j.fertnstert.2017.10.008. Epub 2017 Nov 23. PMID 29175066
- [Background] Armstrong S, Bhide P, Jordan V, Pacey A, Marjoribanks J, Farquhar C. Time-lapse systems for embryo incubation and assessment in assisted reproduction. Cochrane Database Syst Rev. 2019 May 29;5(5):CD011320. doi: 10.1002/14651858.CD011320.pub4. PMID 31140578
- [Background] Kalleas D, McEvoy K, Horne G, Roberts SA, Brison DR. Live birth rate following undisturbed embryo culture at low oxygen in a time-lapse incubator compared to a high-quality benchtop incubator. Hum Fertil (Camb). 2022 Feb;25(1):147-153. doi: 10.1080/14647273.2020.1729423. Epub 2020 Feb 26. PMID 32098536